CLINICAL TRIAL: NCT00724087
Title: Sleep, Energy Metabolism and Diabetes Risk.
Brief Title: Sleep Loss and Energy Metabolism in People With Family History of Type 2 Diabetes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 16079A-S4; R01HL089637 (NIH)
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Sleep; Sleep Deprivation; Insulin Resistance; Type 2 Diabetes
Keywords: short sleep duration; energy expenditure; insulin secretion; insulin action; lipid turnover; free fatty acids
MeSH Terms: conditions — Sleep Deprivation; Insulin Resistance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5.5-hour bedtime (Experimental)
  Interventions: Other: 5.5-hour bedtime
- 8.5-hour bedtime (Experimental)
  Interventions: Other: 8.5-hour bedtime

INTERVENTIONS:
Other: 5.5-hour bedtime — 16 days with sleep allowed only during a 5.5-hour bedtime period at night
  Arms: 5.5-hour bedtime
Other: 8.5-hour bedtime — 16 days with sleep allowed only during a 8.5-hour bedtime period at night
  Arms: 8.5-hour bedtime

SUMMARY:
The use of energy from food changes when people sleep. However, it is still not known if differences in the amount of nighttime sleep have an effect on the amount of energy that people who have a relative with type 2 diabetes (parent, sibling, or grandparent) use to perform their daily activities. This study is being done to test the hypothesis that the daily use of energy in people who have a history of type 2 diabetes in their family will be different after they have slept short hours for 16 days in comparison to when they have slept longer hours for 16 days.

DETAILED DESCRIPTION:
Study participants will complete two 16-day inpatient stays in the sleep laboratory of the University of Chicago Clinical Resource Center that will be scheduled at least 4 weeks apart. Bedtime duration will be set at 5.5 hours per night during one of these stays and at 8.5 hours per night during the other. No daytime naps will be allowed. Study participants will be served regular daily meals including breakfast, lunch, dinner, and a bedtime snack. On weekdays all participants will engage in simulated "office work" in the sleep laboratory. During the rest of the time participants will maintain their usual indoor and outdoor activities as much as possible within the limits of the University of Chicago campus. At the beginning of each inpatient stay, study participants will drink a glass of water containing harmless non-radioactive dense forms of oxygen and hydrogen, small amounts of which are found in natural water. Several urine samples will be collected before and after the participants drink the water and again 14 days later in order to measure the amount of energy that was used by them during this time. At the end of each stay participants will also undergo measurements of their body composition (lean tissue, bone and fat) and their metabolic rate at rest and after a standard meal, and will complete tests to determine how much insulin does their body produce in response to an intravenous glucose infusion and how effective is the action of the sugar-processing hormone, insulin, in their body when it is infused intravenously together with glucose over a period of several hours.

ELIGIBILITY:
Inclusion Criteria:

* regular sleep habits
* BMI 20 to 27 kg/m2
* at least one parent, sibling or grandparent with type 2 diabetes
* must exercise regularly

Exclusion Criteria:

* active smoker
* night or shift work
* have highly variable sleep habits
* have a hormonal disorder
* have a sleep disorder
* have an active medical problem
* women only: use of birth control pills
* women only: irregular menstrual periods or pregnancy
* use of medications/compounds that can disrupt sleep

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Total energy expenditure | during each bedtime intervention

SECONDARY OUTCOMES:
Physical activity related energy expenditure | during each bedtime intervention
Total body insulin sensitivity | at the end of each bedtime intervention
First and second phase insulin secretion | at the end of each bedtime intervention
Endogenous glucose production | at the end of each bedtime intervention
Glycerol turnover and free fatty acid concentration | at the end of each bedtime intervention

CONTACTS AND LOCATIONS:
Overall Officials: Plamen D Penev, MD, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States